CLINICAL TRIAL: NCT04368637
Title: Acute Cardiovascular Events Triggered by COVID-19-Related, Non-infectious Stress The Jordan COVID-9 caRdiovascular Events (JoCORE) Study
Brief Title: Acute Cardiovascular Events Triggered by COVID-19-Related Stress
Acronym: JoCORE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Principal Investigator, Ayman J. Hammoudeh, MD, FACC, Interventional Cardiologist, Jordan Collaborating Cardiology Group
Other Study IDs: JCCG.JoCORE.4.4040
Record Dates: First submitted 2020-04-26; First posted 2020-04-30 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Acute Myocardial Infarction; Ventricular Tachycardia; Sudden Cardiac Death; Stroke, Acute
Keywords: COVID-19; triggered myocardial infarction; triggered acute cardiovascular events; COVID-19-related stress
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac; Stroke; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current COVID19 pandemic has afflicted almost the whole globe. The stress related to the pandemic, not the direct virus-related injury, can be potentially associated with acute cardiovascular events due to a large list of physical and psychosocial stresses.

This study is a cross sectional study that will enroll patients evaluated during the COVID19 pandemic period for acute cardiovascular events.

DETAILED DESCRIPTION:
The onset of acute myocardial infarction (AMI) is a complex interplay of internal circadian factors and external physical and emotional triggers. These interactions may lead to rupture of an often non-occlusive vulnerable atherosclerotic coronary plaque with subsequent formation of an occlusive thrombus. Physical and emotional stresses are important triggers of acute cardiovascular events including AMI. Triggering events, internal changes, and external factors vary among different geographical, environmental, and ethnic regions. Life-style changes, pharmacotherapy, and psychological interventions may potentially modify the response to, and protect against the effects of triggering events. Certain times in the life span of different communities all around the world are prone to natural and man-made disasters that, not only have direct negative impact on human lives and state-resources, but also have indirect impact on triggering acute cardiovascular events during the time of the disaster and the period immediately after. For example, earthquakes, wars, and terrorist attacks, in addition to direct human life loss and destruction of communities, have bees associated with a surge in the number of acute MI, sudden cardiac death, ventricular tachy-arrhythmia and implantable cardiovertor defibrillators (ICD) discharges.

The current COVID-19 pandemic has afflicted almost the whole globe. The virus can directly attack the myocyte and cause various degrees of cardiac damage and cardiovascular clinical entities. However, the stress related to the pandemic, not the direct virus-related injury, can be potentially associated with acute cardiovascular events due to a large list of physical and psycho-social stresses such as extreme physical effort, lock down, anger, fear, financial stress, sorrow, death of a significant person..etc.

This study is a cross sectional study that will enroll patients evaluated during the COVID-19 pandemic period for acute cardiovascular events not directory related to the virus infectivity, who voice certain and specific trigger(s) related to the pandemic impact on social life and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Acute MI (STEMI and NSTEMI).
* Sudden cardiac death
* Ventricular tachycardia
* ICD shocks.
* Stressful trigger prior to the cardiovascular event

Exclusion Criteria:

* COVID-19 infection.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All comers to the ER reporting acute cardiovascular event as pre-specified above. The patient reporting a physical or social stress directly related to the COVID-19 pandemic such as anger, fear, death of a significant person, financial stress, eating binge, extreme physical effort, etc..
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-05-03 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Acute cardiovascular event triggered by COVID-19 stress | 4 months
  Acute myocardial infarction as diagnosed by ST segment elevation or depression or inverted T wave on 12-lead EKG and elevated levels of cardiac troponins above the 99% of the normal values.
  A. Acute MI (STEMI and NSTEMI). B. Aborted on non-aborted sudden cardiac death not attributed to a known etiology.
  C. Sustained or non-sustained ventricular tachy-arrhythmia not attributed to a known etiology.
  D. ICD shocks. 3. Absence of suspected or confirmed infection with the COVID19 virus. 4. Definite physical or psycho-social stressful trigger appearing in relation to the COVID-19 situation (lock down stress, financial stress, anger, depression, fear, sorrow, death of a significant person, eating binges, smoking binges, physical stress [carrying walking for shopping and carrying excess weights] ..etc) as judged by a unanimous agreement of three investigators in the steering committee.
Ventricular tachycardia | 4 months
  Typical ventricular tachycardia on 12-lead EKG or EKG monitor.
acute stroke | 4 months
  acute neurological symptoms of hemiparesis or dysrthria due to brain ischemia proven by computerized tomography or magnatic resonance
Implantable cardioverter defibrillator (ICD) shock | 4 months
  Finding an episode of ventricular tachycardia on interrogation of ICD tracing

CONTACTS AND LOCATIONS:
Overall Officials: Ayman J Hammoudeh, MD, FACC, Study Chair — JCC Group
Locations (5):
- Jordan (5):
  - Istishari Hospital, Amman
  - Abdelhadi Hospital, Amman
  - Farah Hospital, Amman
  - Jordan Hospital, Amman
  - Specialty Hospital, Amman

IPD SHARING:
Plan to Share IPD: No
Baseline clinical data of participating patients will be shared along with the type of the triggered cardiovascular events and the type of trigger implicated in precipitating the event.